CLINICAL TRIAL: NCT03410030
Title: Phase IB/II Trial of High Dose Ascorbic Acid (AA) + Nanoparticle Paclitaxel Protein Bound + Cisplatin + Gemcitabine (AA NABPLAGEM) in Patients Who Have No Prior Therapy for Their Metastatic Pancreatic Cancer
Brief Title: Trial of Ascorbic Acid (AA) + Nanoparticle Paclitaxel Protein Bound + Cisplatin + Gemcitabine (AA NABPLAGEM)
Acronym: AA NABPLAGEM
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: HonorHealth Research Institute (Other)
Collaborators: Stand Up To Cancer (Other); Cancer Research UK (Other); Lustgarten Foundation (Other); Translational Genomics Research Institute (Other); Princeton University (Other); Salk Institute for Biological Studies (Other); Cold Spring Harbor Laboratory (Other); Barts Cancer Institute (Other); University of Arizona (Other); Imaging Endpoints (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU2C HRI NPG-002
Record Dates: First submitted 2018-01-09; First posted 2018-01-25 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Pancreatic Cancer; Pancreas Cancer; Pancreatic Adenocarcinoma Resectable; Pancreatic Ductal Adenocarcinoma; Pancreas Metastases
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Ascorbic Acid; Taxes; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ascorbic Acid (Experimental): Some human studies of high-dose IV vitamin C in patients with cancer have shown improved quality of life, as well as improvements in physical, mental, and emotional functions, symptoms of fatigue, nausea and vomiting, pain, and appetite loss. Intravenous high-dose ascorbic acid has caused very few side effects in clinical trials
  Interventions: Drug: Ascorbic Acid; Drug: Paclitaxel protein-bound; Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Ascorbic Acid — combination therapy
  Other Names: Paclitaxel protein bound; Cisplatin; Gemcitabine
Drug: Paclitaxel protein-bound — combination therapy
  Other Names: Ascorbic Acid; Cisplatin; Gemcitabine
Drug: Cisplatin — combination therapy
  Other Names: Paclitaxel protein-bound; Gemcitabine; Ascorbic Acid
Drug: Gemcitabine — combination therapy
  Other Names: Cisplatin; Paclitaxel protein-bound; Ascorbic Acid

SUMMARY:
The purpose of this study is to see if a treatment regimen with a combination of paclitaxel protein bound (also known as nab-paclitaxel), gemcitabine, and cisplatin when given with high dose Ascorbic Acid will be safe and effective in individuals with untreated metastatic pancreatic cancer.

DETAILED DESCRIPTION:
Pancreatic cancer continues to be a very lethal disease. It was estimated that in 2016, 53,070 Americans would be diagnosed with pancreatic ductal adenocarcinoma (PDA), and 41,780 would die from the disease. This makes pancreatic cancer the third leading cause of death from cancer in the US.

PDA is the twelfth most common cancer in the world with 338,000 new cases diagnosed in 2012. It is estimated that worldwide there will be > 300,000 deaths from pancreatic cancer. Furthermore unfortunately PDA is projected to be the second leading cause of death from cancer in the US by 2030.

Detection of pancreatic cancer has notoriously been very late in the disease and therefore the 5-year survival rate is only 8%, which is actually a slight improvement over the last few years. Right now the only potential cure for pancreatic cancer is surgical resection (if the disease is caught early). However only about 20% of PDA patients are eligible for potentially curable resection and unfortunately most (> 80%) have recurrence of their cancer within 2 years of resection, and those recurrences are almost universally fatal.

Recently it has been shown that there are regimens that actually improve survival for patients with advanced stage IV PDA. Conroy and colleagues have developed the Folfirinox regimen, which in a large randomized trial improved survival over gemcitabine as a single agent. Von Hoff and colleagues developed the nanoparticle albumin (nab) associated paclitaxel plus gemcitabine regimen which improved survival over single agent gemcitabine. Even more recently Jameson and colleagues have presented a combined regimen of nab-paclitaxel + gemcitabine + cisplatin in a small 24 patient phase Ib/II trial which showed a response rate of 71% with 2 patients having complete response, a 1-year survival of 65% and a median survival of 16+ months.

While there have been multiple investigators and investigations into the use of ascorbic acid for patients with cancer (see ClinTrials.gov), its use has generally not been found to be of help for patients particularly when given orally - e.g. 10 grams daily.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria to be included in the trial:

* Be willing and able to provide written informed consent/assent for the trial.
* Be ≥ 18 years of age on day of signing informed consent.
* Histologically or cytologically confirmed metastatic pancreatic adenocarcinoma (with measurable disease according to RECIST 1.1 criteria).
* Have a performance status of 0 or 1 on the ECOG performance scale.
* Demonstrate adequate organ function as defined below in table 4. All screening labs should be performed within 14 days of treatment initiation.
* Female participants of childbearing potential should have a negative serum pregnancy test within 72 hours prior to receiving first dose of study medication.
* Female participants of childbearing potential must be willing to use adequate method of contraception (as outlined in section 4.4.2) for the duration of the trial.
* Male participants must agree to use adequate contraception (as outlined in section 4.4.2) for the duration of the trial.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the participant.

Exclusion Criteria:

Patients must not meet any of the following criteria in order to be eligible for the trial:

* Patients must have received no previous radiotherapy, surgery, chemotherapy or investigational therapy for the treatment of metastatic disease. Prior treatments in the adjuvant setting with gemcitabine and/or 5-FU or gemcitabine administered as a radiation sensitizer are allowed, provided at least 6 months have elapsed since completion of the last dose and no lingering toxicities are present.
* Palliative surgery and/or radiation treatment less than 4 weeks prior to initiation of study treatment.
* Exposure to any investigational agent within 4 weeks prior to initiation of study treatment.
* Patients who need constant use of finger stick blood glucose monitoring for tight contro l of their diabetes being the ascorbic acid causes false low readings of glucose via that technology (Vasudevan and Hirsch 2014) 39
* Any person with a G6PD deficiency
* History of renal oxalate stones (if type of stone is unknown, need to assess urine oxalates level if >60mg/dL, then patient is not eligible for the study)
* Patient is taking acetaminophen at any dose, or any medication that contains acetaminophen within 72 hours of first dose of ascorbic acid.
* Hypersensitivity to any of the agents proposed for treatment.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through one week from the last dose of trial treatment.
* Patients with evidence of iron overload, defined as a transferrin saturation > 45 percent AND serum ferritin > 200 ng/mL (males) or >150 ng/mL (females).
* Current, serious, clinically significant cardiac arrhythmias as determined by the investigator, or patient receiving a digitalis derivative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Phase IB: Recommended Phase II dose (to give ≥ 20 mM) of ascorbic acid for Phase II | approximately 63 days
  To determine the maximum tolerated dose (MTD) of high dose ascorbic acid (AA) with triple therapy of nanoparticle paclitaxel protein bound+ cisplatin + gemcitabine (NABPLAGEM) in patients with advanced stage IV metastatic pancreatic cancer
Phase II: Disease control rate (CR+PR+SD x18 weeks) | approximately 63 days
  To determine the preliminary efficacy (Disease control rate of CR+ PR+SD X 18 weeks) of the combination of high dose ascorbic acid (AA) at MTD with triple therapy of nanoparticle albumin- bound paclitaxel + cisplatin + gemcitabine (NABPLAGEM) in patients with advanced stage IV metastatic pancreatic cancer.

SECONDARY OUTCOMES:
Incidence of toxicities | approximately 63 days
  Lab testing will be completed to evaluate standard of care labs for subject safety
Percent of patients who normalize their CA19-9 | approximately 63 days
  Lab testing will be completed to evaluate normalization of CA19-19
overall survival | approximately 12 weeks from last study treatment
  Telephone followup will be conducted every 12 weeks from the last dose of treatment to determine survival status
Progression free | approximately 12 weeks from last study treatment
  Telephone followup will be conducted every 12 weeks from the last dose of treatment to determine status of disease progression
Changes in patient's self-reported quality of life | approximately 63 days
  Changes in patient's self-reported quality of life will be determined by administering the MD Anderson Symptom Inventory (MDASI-GI)
Changes in patient's self-reported pain levels | approximately 63 days
  Changes in patient's self-reported pain levels will be determined by administering the Brief Pain Inventory (BPI)

OTHER OUTCOMES:
Tumor texture on radiologic scans | approximately 63 days
  Imaging will be completed to evaluate tumor texture on radiologic scans as a non-invasive imaging biomarker for response, biologic, pathologic and outcome measures
Correlation between peak plasma concentration of ascorbic acid and response to treatment | approximately 63 days
  Lab testing will be completed to evaluate the correlation between peak plasma concentration of ascorbic acid and response to treatment
Potential tumor biomarkers | approximately 63 days
  Tumor biopsy testing will be completed to evaluate potential biomarkers in the tumor including tumor immune cell infiltration, stromal activation, stem cell enumeration, metabolic profiles, whole exome and whole genome CN, ChIP-seq/ATAQ seq, IHC and PCR assays on immune cell populations, CAFs, stem cell content (CD133, Aldh) and Musashi
Potential blood biomarkers | approximately 63 days
  Lab testing will be completed to evaluate potential biomarkers in the blood samples. Test may include CTCs/circCSC enumeration, Single CTC/circCSC transcription profiling, immune profiling [CD4+CD8+ T cells, MDSC (IDO-1+HLR-DR-/lowCD33+CD11b+CD14+), Immunosuppressive plasmocytes (CD19+CD138+IgA+IL-10+PD-L1+), Th17 (CD3+gdTCR+IL-17A+), Treg (CD4+Foxp3+), Hypo-responsive NK cells (CD3-CD56+KIR-NKG2A-), cfDNA, GPC1+ exosomes.
Changes in circulating tumor stem cells | approximately 63 days
  Lab testing will be completed to evaluate changes in numbers of circulating tumor stem cells and macrophage lineage changes

CONTACTS AND LOCATIONS:
Overall Officials: Gayle S Jameson, RN, MSN, ACNP-BC, AOCN, Principal Investigator — HonorHealth Research Institute
Locations (1):
- HonorHealth Research Institute, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
If the study site is a 'covered site' under the definitions of the Health Insurance Portability and Accounting Act (HIPAA), the Investigator will ensure that the patient consents to the use of data by HonorHealth and its designees for the purposes of regulatory submissions, study publications, and drug approval.
  SU2C will be notified of any outputs of the research such as guidelines, publications, presentation, changes in service delivery etc. prior to external submission or presentation. In any oral or written report or poster presentation of Results or otherwise relating to the Research, the support of CRUK, SU2C and the Lustgarten foundation will be acknowledged, displaying the relevant logs where possible. Any publications resulting from research funded in whole or in part by the Grant must be cited as required per signed confidentiality agreements.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: to be determined
Access Criteria: The Investigator and any other study personnel involved in this study shall not disclose, or use for any purposes (other than for the performance of this study), any data, records, or other information (hereinafter collectively "information") disclosed to the Investigator or other study personnel. Such information shall remain the confidential and proprietary property of HonorHealth, and shall be disclosed only to the Investigator or other designated study personnel.
  The obligation of non-disclosure shall not apply to the following:
  * relevant disclosure to potential study participants for the purpose of obtaining informed consent;
  * information after such time that it is or becomes publicly available through no fault of the Investigator or other study personnel; and,
  * information after such time that it is disclosed to the Investigator by a third party entitled to disclose such information.

REFERENCES:
- [Derived] Jameson GS, LeGrand SD, Gordon MS, Roe DJ, Wertheim BC, Olszewski K, Rabinowitz J, Evans R, Downes M, Truitt M, Korn R, Han H, Miller RM, Barrett MT, Propper D, Von Hoff DD, Borazanci E. Phase IB trial of high dose ascorbic acid + nab-paclitaxel + cisplatin + gemcitabine in patients with untreated metastatic pancreatic cancer. Redox Biol. 2025 Dec;88:103895. doi: 10.1016/j.redox.2025.103895. Epub 2025 Oct 25. PMID 41197185